CLINICAL TRIAL: NCT02476539
Title: An Ascending Single and Multiple Dose Study of the Pharmacokinetics, Safety and Tolerability of the Irreversible Epidermal Growth Factor Receptor Inhibitor Hemay022 in Patients With HER2-Positive Advanced Breast Cancer
Brief Title: Study Evaluating Hemay022 In Subjects With HER2-Positive Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hemay022-002
Record Dates: First submitted 2015-06-11; First posted 2015-06-19 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: HER2 Positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemay022 (Experimental): Part one: Dose Escalation Group Hemay022 tablets will be taken orally once daily in doses of 50mg, 100mg, 200mg, 300mg,400mg or 500mg daily for 28 days.
  Part two: Extension Group Hemay022 tablets will be taken in three dose groups that had been assessed by Part one for 28 days.
  Interventions: Drug: Hemay022

INTERVENTIONS:
Drug: Hemay022

SUMMARY:
The purposes of this study are to assess the safety, tolerability and pharmacokinetics of Hemay022. The secondary purpose of this study is to assess the efficacy of Hemay022 in the treatment of HER2-positive advanced breast cancer.

The study will be conducted in two parts. Part one, trial will be conducted in 18-30 subjects to determine safety and tolerability of Hemay022 in patients with HER2-positive advanced breast cancer. Part two, approximately 27 additional subjects with HER2-positive advanced breast cancer, are included to better define the tolerability and preliminary efficacy of Hemay022.

DETAILED DESCRIPTION:
This is a phaseⅠsequential-group study of ascending single and multiple oral doses administered to subjects with HER2-Positive Advanced Breast Cancer. Each subject will receive a single dose of Hemay022, followed by a 1-week observation period, and then will receive Hemay022 administered once daily by mouth for 28 days. Each cycle consist of 28 days. Subjects will be enrolled in groups of 3 to 6. Depending on the safety and activity profile observed during the dose escalation phase, the dose selected for Part 2 may be adjusted. Part 2 is an extension part of three dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 65 years;
2. Histologically or cytologically confirmed and radiologically diagnosed advanced breast cancer subjects; and subjects who have failed standard therapy，or no effective therapy available for such subjects
3. HER2 over-expression by IHC with score of 3+, or 2+ with FISH confirmation;
4. Preferably measurable tumour lesion as defined by RECIST criteria1.1;
5. Subjects have received chemotherapy at least 4 weeks prior to screening (at least 6 weeks of washout time frame if treated with mitomycin and nitrosoureas) and must have recovered from any toxic effects of the treatment --- to CTCAE 4.03≤ Grade 1;
6. ECOG Performance Status of 0,1;
7. Life expectancy of at least three months;
8. Adequate bone marrow, liver, kidney function, meeting the following creteria:

   ANC≥1.5×109/L, HB≥90g/L, PLT≥75×109/L； TBIL≤1.5×ULN, ALT≤1.5×ULN, AST≤1.5×ULN; Cr ≤1×ULN; BUN ≤1×ULN;
9. Left ventricular ejection fraction (LVEF) ≧50% as measured by Ultrasonic cardiogram (UCG)
10. All female and male subjects must agree and commit to the use of a reliable contraceptive regimen for the duration of the study and for at least 12 weeks after at the last dose of test article. Female subjects must have a negative serum or urine pregnancy test performed within 7 days prior to treatment;
11. Ability to understand and the be willingness to sign a written informed consent before study entry;
12. subjects would have good communication with the investigator and could comply with protocol

Exclusion Criteria:

1. Patients with parenteral nutrition; malabsorption syndrome; or any condition possibly affecting drug absorption or inability to tolerate oral medications;
2. Clinically QTc prolongation, ventricular tachycardia, ventricular fibrillation, heart block, myocardial infarction within 1 year, congestive heart failure, symptoms requiring medicine treatment patients with coronary heart disease;
3. Ventricular ejection fraction (LVEF) <50％;
4. Active infection (ie, requiring intravenous antibiotic or antiviral agent);
5. Active central nervous system metastases
6. Have received other clinical trials treatment within the 4 weeks prior to study;
7. Have received other target therapy within the 4 weeks prior to study;
8. Pregnant or breast feeding women;
9. Have a known hypersensitivity to the test article or any of the excipient of the test article;
10. Evidence of significant medical illness or abnormal laboratory finding that would make the subject inappropriate for this study by the investigator's judgment.
11. Subjects cannot complete the study due to other reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 4 weeks of treatment
Observed maximum concentration of Hemay022 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on day 1 and day 35
Time of maximum concentration of Hemay022 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on day 1 and day 35
Area under the plasma concentration versus time curve of Hemay022 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on day 1 and day 35
Trough Plasma Concentrations of Hemay022 | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on day 1 and day 35
Predose plasma concentration | Predose on day 7, 14, 21

SECONDARY OUTCOMES:
Disease control rate (complete response rate + partial response rate + stable disease rate) according to RECIST v1.1 | 4 weeks of treatment
Objective response rate (complete response rate + partial response rate) according to RECIST v1.1 | 4 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China